CLINICAL TRIAL: NCT03428321
Title: Small and Steatotic Hepatocellular Carcinoma : a Distinctive Radiological Variant With Improved Outcome After Percutenous Ablation
Brief Title: Small and Steatotic Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0436
Record Dates: First submitted 2018-01-08; First posted 2018-02-09 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: HCC
Keywords: Microwave ablation; Percutaneous thermalablation; High risk location; Articifial pneumothorax; Lipiodol marked; Prognostic factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous thermoablation in an effective local curative treatment in patients with cirrhosis and HCC smaller than 3 cm in diameter (BCLC 0-A).

Around 30% of HCC patients referred for percutaneous ablation were regarded as non-feasible because of a difficult-at risk location or undetectable nodules.

We used percutaneous thermoablation to treat HCC on high risk locations (subcapsular or liver dome) with or without lipiodol marked (for undetectable HCC).

No clinical study has been published so far to compare percutaneous thermoablation of HCC on liver dome CT guided with artificial pneumothorax and lipiodol marked, and percutaneous thermoablation of HCC guided by ultrasonography (non subcapsular, distent form diaphragm).

This retrospective study evaluate the overall survival, the local tumor progression or distant liver progression after percutaneous ablation for HCC and determine prognostic factors.

DETAILED DESCRIPTION:
We performed 412 percutaneous thermoablations on 238 patients for HCC between January 2015 and November 2019.

All thermoablation procedures were performed percutaneously under ultrasound or CT guidance, with ou without artificial pneumothorax or ascites, with ou without lipiodol marked.

Purposes:

* Tumor response upon mRECIST criteria
* Progression-free survival
* Overall survival
* Local tumor progression
* Distent liver progression
* Prognostic factors

ELIGIBILITY:
Inclusion criteria:

* HCC according to histological examination or Barcelona criteria
* BCLC0 or A
* Measurable targets according to mRECIST v1.1
* Child A or B7 cirrhosis
* HCC < 4 cm, < 3 nodules, Age ≥ 18 years
* No extrahepatic metastasis, no vascular invasion
* Performance status 0 or 1
* Thrombocytes ≥ 50 000/mm3, TP > 50%

Exclusion criteria:

* Follow-up < 1month
* Lobar/main portal venous thrombus
* Abundant ascites
* Antecedent of bilio-digestive anastomosis or endoscopic sphincterotomy
* Combined treatment with embolization or chemo-embolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent one or several percutaneous thermoablations for HCC form January 2015 to November 2019 at the Department of Radiology St-Eloi University Hospital - Montpellier School of Medicine France.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Thermal ablations | 1 day
  Evaluation of thermal ablations (radiofrequency and microwave ablation)

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC